CLINICAL TRIAL: NCT06423209
Title: Efficacy of an Omnivorous Versus a Vegan Diet in the Prevention or Treatment of Sarcopenia in Chilean Adults Following a Strength Training Program
Brief Title: Efficacy of a Training Program in Adults Following a Vegan Diet Versus an Omnivorous Diet
Acronym: Vegan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Concepcion (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CEBB 1068-2021
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Physical Activity
Keywords: vegan diet; omnivorous diet; strength training
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: The study consisted of a 4-arm non-randomized controlled clinical trial, with measurements at the beginning and end of a 16-week intervention.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Vegan Intervention (Experimental): The intervention group is composed of people who follow a vegan diet and who will be part of an intervention program for 16 weeks, consisting of a physical exercise program of strength resistance with 3 sessions per week. Each session will be guided by a physical activity professional and will last from 45 to 50 minutes.
  Interventions: Other: Strength training program
- omnivorous intervention (Experimental): The intervention group is composed of people who follow a omnivorous diet and who will be part of an intervention program for 16 weeks, consisting of a physical exercise program of strength resistance with 3 sessions per week. Each session will be guided by a physical activity professional and will last from 45 to 50 minutes.
  Interventions: Other: Strength training program
- vegan control (No Intervention): People who follow an vegan diet who were part of the control group. They were evaluated before and after the intervention.
- omnivorous control (No Intervention): People who follow an omnivorous diet who were part of the control group. They were evaluated before and after the intervention.

INTERVENTIONS:
Other: Strength training program — Strength training program to be developed during 16 weeks. There will be 3 exercise sessions per week and those participants who perform at least 2 sessions during the program will be considered for the statistical analysis.
  Arms: Vegan Intervention; omnivorous intervention

SUMMARY:
The study consisted of a non-randomized controlled clinical trial with measurements at baseline and at the end of a 16 week intervention. Participants will be assigned to the intervention or control group according to their own choice and convenience. A 4 arm split was performed where the Veg-Int group was composed of people on a vegan diet who participated in the intervention, the Veg-Con group was composed of people on a vegan diet who were part of the control group, the Omn-Int group was composed of people on an omnivorous diet who participated in the intervention, and the Omn-Con group was composed of people on an omnivorous diet who were part of the control group.

The Veg-Int and Omn-Int intervention groups, participated in a physical exercise program in remote modality through a digital mHealth platform. During the 16 weeks of intervention, a total of 50 training sessions were carried out, distributed in three sessions per week, with a duration per session ranging from 40 to 50 minutes. The exercise program was designed and supervised by a physical education teacher and focused on strength training using body weight exercises targeting the major muscle groups, including upper body, lower body and abdominals. The platform recorded participants attendance and the time they spent on each exercise session. At the end of the sessions, participants had the option to evaluate and share their perception of effort during the workout through a Modified Borg scale (0-10). In addition, they were given the opportunity to communicate with the teacher via phone call, text message or e-mail, to receive feedback or raise doubts.

DETAILED DESCRIPTION:
All participants were evaluated in weeks 0 and 17, immediately after the intervention program, under the same conditions in terms of protocol, calibrated instruments and the same evaluator.

The evaluation of nutritional status was carried out using the body mass index (BMI, Kg/m2), while the waist circumference was measured by passing a measuring tape at the height of the navel, midpoint between the costal margin and the crest. iliac, at the end of a normal expiration and recorded in centimeters.

Body composition analysis was obtained by the bioimpedance method, using a segmented bioimpedance meter. The measurements were carried out under fasting conditions for at least 4 hours, without having performed physical exercise in the last 12 hours, without consuming stimulating drinks such as caffeine and avoiding the menstrual period. From the body composition information, the data Percentage of Fat Mass, Kilos of Fat Mass and Kilos of Lean Mass were recorded.

The level of physical activity was assessed through a self-report questionnaire of physical activity and sitting time in the last 7 days, using the abbreviated version of the International Physical Activity Questionnaire (. The questionnaire was administered by a physical activity professional, and the data were reported in minutes per day to estimate the total PA performed, and the time reported was corrected by its metabolic equivalent .

The type of diet was corroborated through a quantified food consumption trend survey, which included 14 groups; vegetables, fruits, dairy and vegetable options, meat-fish-seafood and egg, legumes, vegan protein preparations, grains and cereals, fats and oils, nuts, sugars and sweets, alcohol, snacks, coffee and infusions, food supplements. The questionnaire was administered individually by a dietitian nutritionist to each participant.

ELIGIBILITY:
Inclusion Criteria:People between 18 and 59 years old who follow a vegan or omnivorous diet for at least the last 6 months prior to the study.

- Exclusion Criteria: Those who were doing strength training or doing less than 3 hours of vigorous exercise per week did not have health compatible with the activities of this study. People with a diagnosis of diabetes, uncontrolled hypertension (Systolic Blood Pressure ≥150 and/or Diastolic Blood Pressure ≥90 mmHg). People who were undergoing treatment for cancer, chronic kidney failure, or who reported a health problem in the previous fitness for physical activity questionnaire (PAR-Q).

-

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2022-02-02 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Body weight | 16 weeks of intervention
  Differential between kg of body weight before and after the development of the intervention
waist circumference | 16 weeks of intervention
  Differential between centimeters of waist circumference before and after the development of the intervention
fat mass | 16 weeks of intervention
  Differential of the percentage of fat mass before and after the intervention
Lean mass | 16 weeks of intervention
  Differential of kilograms of lean mass before and after the intervention
maximum strength | 16 weeks of intervention
  Differential of kilograms of maximum strength by biceps curl exercise
Manual grip strength | 16 weeks of intervention
  Differential of manual grip strength of both hands using a hydraulic dynamometer.
Vertical jump | 16 weeks of intervention
  Differential evaluation of muscle power by means of a vertical jump

CONTACTS AND LOCATIONS:
Overall Officials: Rafael E Zapata Lamana, Doctor, Study Director — Universidad de Concepcion
Locations (1):
- Richar Carcamo Regla, Concepción, Concepcion, Chile

IPD SHARING:
Plan to Share IPD: No
Has not been considered or discussed yet

REFERENCES:
- [Background] Boutros GH, Landry-Duval MA, Garzon M, Karelis AD. Is a vegan diet detrimental to endurance and muscle strength? Eur J Clin Nutr. 2020 Nov;74(11):1550-1555. doi: 10.1038/s41430-020-0639-y. Epub 2020 Apr 24. PMID 32332862
- [Background] Hevia-Larrain V, Gualano B, Longobardi I, Gil S, Fernandes AL, Costa LAR, Pereira RMR, Artioli GG, Phillips SM, Roschel H. High-Protein Plant-Based Diet Versus a Protein-Matched Omnivorous Diet to Support Resistance Training Adaptations: A Comparison Between Habitual Vegans and Omnivores. Sports Med. 2021 Jun;51(6):1317-1330. doi: 10.1007/s40279-021-01434-9. Epub 2021 Feb 18. PMID 33599941
- [Background] Reid-McCann RJ, Brennan SF, McKinley MC, McEvoy CT. The effect of animal versus plant protein on muscle mass, muscle strength, physical performance and sarcopenia in adults: protocol for a systematic review. Syst Rev. 2022 Apr 13;11(1):64. doi: 10.1186/s13643-022-01951-2. PMID 35418173
- [Background] van de Brekel JA, Duurkens VA, Vanderschueren RG. Pneumothorax. Results of thoracoscopy and pleurodesis with talc poudrage and thoracotomy. Chest. 1993 Feb;103(2):345-7. doi: 10.1378/chest.103.2.345. PMID 8432116
- [Background] Hannaian SJ, Churchward-Venne TA. Meatless Muscle Growth: Building Muscle Size and Strength on a Mycoprotein-Rich Vegan Diet. J Nutr. 2023 Jun;153(6):1665-1667. doi: 10.1016/j.tjnut.2023.04.011. Epub 2023 Apr 14. No abstract available. PMID 37062484
- [Background] Pohl A, Schunemann F, Bersiner K, Gehlert S. The Impact of Vegan and Vegetarian Diets on Physical Performance and Molecular Signaling in Skeletal Muscle. Nutrients. 2021 Oct 29;13(11):3884. doi: 10.3390/nu13113884. PMID 34836139